CLINICAL TRIAL: NCT04083729
Title: Predictors of Persistent Pulmonary Hypertension After Percutaneous Mitral Commissurotomy and Its Impact on Clinical Outcomes
Brief Title: Persistent Pulmonary Hypertension After Percutaneous Mitral Commissurotomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Abdel Fattah Mohamed Ahmed, Assistant Lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PH after mitral commissurtomy
Record Dates: First submitted 2019-08-29; First posted 2019-09-10 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Intervention Model Description: predictors of Persistent Pulmonary Hypertension After Percutaneous Mitral Commissurotomy
Who Masked: Participant
Masking Description: percutaneous mitral commissurotomy
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with persistent pulmonary hypertension (Active Comparator): Patients with persistent pulmonary hypertension after balloon mitral comisseruotomy
  Interventions: Procedure: Percutaneous Mitral Commissurotomy
- Patients without persistent pulmonary hypertension (Active Comparator): Patients without persistent pulmonary hypertension after balloon mitral comisseruotomy
  Interventions: Procedure: Percutaneous Mitral Commissurotomy

INTERVENTIONS:
Procedure: Percutaneous Mitral Commissurotomy — Percutaneous mitral commissurotomy is performed by experienced interventional cardiologists using the Inoue balloon or multitrack technique. During the procedure, conventional hemodynamic parameters are monitored. A successful immediate result is defined as a mitral valve area > 1.5 square cm with less than moderate to severe mitral regurgitation.
  Other Names: Percutaneous mitral valvuloplasty

SUMMARY:
To identify clinical, echocardiographic, and hemodynamic parameters which can predict persistent PH after PMC, and also to determine the impact of persistent PH on the clinical outcomes.

DETAILED DESCRIPTION:
Pure mitral Stenosis develops in approximately 40% of all patients with rheumatic heart disease, and is frequently complicated by Pulmonary hypertension (PH). Pulmonary hypertension influences symptomatology and long-term prognosis. Percutaneous Mitral Commissurotomy (PMC), was first described in 1984, has good results and is performed by antegrade access to the mitral valve through trans-septal puncture by one of various techniques (e.g. Inuoe, and multitrack system). Pulmonary artery pressures (PAP) decrease following PMC. The improvement in pulmonary hypertension after PMC is explained by the improvement in the mitral valve area and subsequent decompression of left atrium (LA) and pulmonary venous beds. Even though there have been studies showing excellent results following PMC in all grades of PH, nonregression of PH following PMC is not uncommon. The component of PAP contributed by the passive transmission of the elevated LA pressure regresses immediately after a successful PMC proportional to the reduction in transmitral gradient. The PH contributed by pulmonary arteriolar constriction slowly comes down over weeks or a few months, But a "fixed" component due to pulmonary vascular disease usually persists.

ELIGIBILITY:
Inclusion Criteria:

* Severe mitral stenosis (mitral valve area ≤1.5cm).
* Significant dyspnea.
* Favorable anatomical characteristics for PMC as assessed by transthoracic echocardiography

Exclusion Criteria:

* Significant mitral regurgitation (≥ grade II/IV). Bilateral commissural calcification.
* Presence of other lesions which need open heart surgery.
* Wilkins' score > 12.
* Persistent LA thrombus despite adequate anticoagulation.
* End stage renal or liver disease.
* Patients with severe COPD and other chest problems that might be complicated by pulmonary hypertension per se.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2019-09 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Composite of cardiovascular event | Participants will be followed for a minimum follow-up of one month
  Composite of cardiovascular mortality, cerebral infarction, systemic embolic events ,RV failure ,MV re stenosis that occurred during follow-up, and PMC-related complications; procedural mortality and urgent MV surgery. parameters changes from base line study and after follow up as MVA in cm 2,PASP in mmHg,LAP in mmHg,LVEP in mmHg,PVR in wood unit

CONTACTS AND LOCATIONS:
Overall Officials: mohamed Abdelghany Koreim, Principal Investigator — Assiut University, 71515 Assiut, Egypt.; Hosam Hasan El Araby, Study Director — Assiut University, 71515 Assiut, Egypt.; Amr ElBadry Ibrahim, Principal Investigator — Assiut University, 71515 Assiut, Egypt.

REFERENCES:
- [Background] Hart SA, Krasuski RA, Wang A, Kisslo K, Harrison JK, Bashore TM. Pulmonary hypertension and elevated transpulmonary gradient in patients with mitral stenosis. J Heart Valve Dis. 2010 Nov;19(6):708-15. PMID 21214093
- [Background] Noor A, Saghir T, Zaman KS. Determinants of decrease in pulmonary hypertension following percutaneous transvenous mitral commissurotomy. J Coll Physicians Surg Pak. 2009 Feb;19(2):81-5. PMID 19208309
- [Background] Bahl VK, Chandra S, Talwar KK, Kaul U, Sharma S, Wasir HS. Balloon mitral valvotomy in patients with systemic and suprasystemic pulmonary artery pressures. Cathet Cardiovasc Diagn. 1995 Nov;36(3):211-5. doi: 10.1002/ccd.1810360304. PMID 8542626
- [Background] Fawzy ME, Osman A, Nambiar V, Nowayhed O, El DA, Badr A, Canver CC. Immediate and long-term results of mitral balloon valvuloplasty in patients with severe pulmonary hypertension. J Heart Valve Dis. 2008 Sep;17(5):485-91. PMID 18980082